CLINICAL TRIAL: NCT05583968
Title: Evaluation of the Efficiency and Accuracy of Artrya-Salix AI Software in the Reporting of Coronary Computed Tomography Angiography Scans in a Real-world NHS Setting. A Retrospective Study.
Brief Title: Efficiency of AI Reporting (EAIR).
Acronym: EAIR
Status: Withdrawn | Type: Observational
Why Stopped: sponsor decision
Sponsor: London North West Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CRC/2021/003
Record Dates: First submitted 2022-05-30; First posted 2022-10-18 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Coronary Artery Disease
Keywords: Artificial Intelligence; Coronary Artery Disease; CCTA; atherosclerotic plaque; vulnerable plaque
MeSH Terms: conditions — Coronary Artery Disease; Plaque, Atherosclerotic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
While there are features on a CCTA that are correlated with plaque vulnerability and can be reported on, this is not always done. This is important as it is thought that vulnerable plaques present the greatest risk of myocardial infarction. This study will assess the correlation between software and human classification of these plaques, as well as demonstrating the time efficiency of AI reporting when compared to a clinician.

DETAILED DESCRIPTION:
This is a retrospective observational study. It will be performed at London Northwest Healthcare NHS Trust (LNWH -Northwick Park Hospital (NPH), Harrow and Ealing Hospital, Southall).

Patients who have had a CCTA in the last 12 months will be contacted about the study. Their CCTA scans will already have been reported and the patient aware of the results. After giving informed consent, 100 patients will have their clinical CCTA images uploaded to the Artrya Salix software for analysis. Simultaneously the images will be re-reported by the physician as per standard of care. Both reports will be obtained and any differences noted. The time the images are sent to Artrya Salix and report received will be recorded. The time the clinician opens the image to analyse and the time when the report is complete will also be recorded using a stopwatch. All images will be analysed by both expert readers to take account of inter-observer variability. The first 30 patients will be treated as a pilot for the study and after their recruitment and image upload and analysis, the team will meet to discuss any issues that have arisen.

During the analysis, any patient who has plaque identified by the software or expert reader will have further analysis of their images. This is to look at the plaques in detail and to compare the sensitivity and specificity of the expert reader analysis. The time it takes for the clinician to report the scans on this group of patients will also be recorded. In addition, assessment will be made of the plaques using comparison of stenosis to calcium score.

.

Data that will be collected will include:

1. Demographic data (age, gender, ethnicity)
2. CCTA results - standard of care
3. CCTA results - Artrya Salix
4. Time from image upload to Artrya Salix to time report received from Artrya Salix
5. Time clinician takes to analyse scan
6. Clinical assessment of plaque for vulnerable characteristics.

The data will be from the electronic medical records of LNWUH NHS Trust. A level 2 or level 3 Cardiology imaging or Radiology Consultant will report the CCTA images.

Data will be captured on an eCRF. The time of image upload to Artrya Salix will be recorded by the system and transposed directly into the eCRF. The time starting and ending image analysis by the clinician will be recorded on a worksheet as source documentation and then entered into the eCRF. A score will be given by the physician as to the likelihood of a plaque being vulnerable where 1= unlikely and 5 = highly likely.

ELIGIBILITY:
Inclusion Criteria:

* Clinical CCTA
* Able to provide informed consent

Exclusion Criteria:

* Unable / unwilling to give informed consent
* Previous CABG or stent insertion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have been referred for CCTA over the last 12 months will be invited to take part. The rationale is to test this software in a real-world setting and this method will provide a non-selective sample. No patient will be contacted until their vital status has been checked on the national SPINE database.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2025-02-09 (Estimated); Study Completion 2025-03-09 (Estimated)

PRIMARY OUTCOMES:
Speed of reporting | Through study completion, up to 26 weeks
  1. Time taken for Artrya Salix reporting of a CCTA scan is as fast or faster than clinician reporting
Vulnerable plaque identification | Through study completion, up to 26 weeks
  2. In a subset of patients where the software has identified vulnerable plaques, this is in agreement with the expert clinical report.

SECONDARY OUTCOMES:
Speed assessing plaque vulnerability | Through study completion, up to 26 weeks
  The secondary outcome of this study will be the additional time taken by the clinician to report plaque vulnerability characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Navtej Chahal, PhD FESC, Principal Investigator — LNWUH NHS Trust
Locations (1):
- London North West University Healthcare NHS Trust, Harrow, Middx, United Kingdom

IPD SHARING:
Plan to Share IPD: No
dat will be fully anonymous and will remain within the study team.